CLINICAL TRIAL: NCT06783075
Title: Milk Vs Wheat Protein Intake to Maximize Whole-body Protein Synthesis Rates in Healthy Older Adults
Acronym: Plant-IAAO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: METC 24-051
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Protein Metabolism
Keywords: whole-body protein synthesis
MeSH Terms: interventions — Milk

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, parallel study design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Protein beverages with milk- or wheat composition will look similar.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MILK (Active Comparator): Drink containing amino acid composition of milk protein
  Interventions: Other: MILK
- WHEAT (Active Comparator): Drink containing amino acid composition of wheat protein
  Interventions: Other: WHEAT

INTERVENTIONS:
Other: MILK — Drink containing amino acids in the composition of milk protein
  Arms: MILK
Other: WHEAT — Drink containing amino acids in the composition of wheat protein
  Arms: WHEAT

SUMMARY:
Dietary protein intake is essential for tissue renewal and growth. Current recommendations for protein intake are based on studies using egg protein as reference protein. Egg protein is an animal-based protein with a high quality. Protein quality is determined by the composition of (essential) amino acids and digestibility. Therefore, different proteins have a different quality. Due to the environmental crisis, an increasing number of people consumes more plant-based proteins. These plant-based proteins often have a lower protein quality compared to animal-based proteins. Therefore, the aim of this study is to investigate whether optimal protein intake depend on protein quality. The optimal protein intake of an animal-based protein with a high quality (milk) will be compared to the optimal protein intake of a plant-based protein with a low quality (wheat).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 65-85 years
* BMI between 18.5-30 kg*m^-2
* Healthy, recreationally active (maximal one intensive exercise training per week)
* No physical limitations (i.e., able to perform all activities associated with daily living independently)

Exclusion Criteria:

* Smoking
* Diagnosed musculoskeletal disorders
* Use of any medications known to affect protein metabolism (i.e., corticosteriods, non-steroidal anti-inflammatories)
* Chronic use of gastic acid-suppressing medication or anti-coagulants
* Unstable weight over the last 3 months
* Diagnosed GI tract disorders or diseases
* Blood donation in the past 2 months

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Differences in protein intake to maximize whole-body protein synthesis rates in older adults based on consumption of milk protein or wheat protein | From enrollment to the end of the study at 7 weeks

SECONDARY OUTCOMES:
Estimated Average Requirement (EAR) to maximize whole-body protein synthesis rates in healthy older adults based on milk protein | From enrollment to the end of the study at 7 weeks
The Recommended Daily Allowance (RDA) to maximize whole-body protein synthesis rates in older adults based on milk protein | From enrollment to the end of the study at 7 weeks
The Estimated Average Requirement (EAR) to maximize whole-body protein synthesis rates in older adults based on wheat protein | From enrollment to the end of the study at 7 weeks
The Recommended Daily Allowance (RDA) to maximize whole-body protein synthesis rates in older adults based on wheat protein | From enrollment to the end of the study at 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon request